CLINICAL TRIAL: NCT00697021
Title: Thromboelastography As An Assessment Tool for Possible Clopidogrel and Aspirin Resistance in The Patients Treated With Primary PCI for STEMI
Brief Title: Thromboelastography As An Assessment Tool for Possible Clopidogrel and Aspirin Resistance
Acronym: TEG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Alex Blatt MD, Intensive Coronary Care Unit Assaf Harofeh MC
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 57/08
Record Dates: First submitted 2008-06-10; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-04

CONDITIONS: Acute ST SEgment Elevation Myocardial Infarction
Keywords: Thromboelastography; Aspirin; Clopidogrel; Plavix; Resistance; Platelet; Coronary Stenting; Bare Metal Stent; Dual antiplatelet therapy; Overreactivity; Primary Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients who suffered acute STEMI and were treated by PPCI and by Aspirin 100mg and Plavix 75mg and showed on treatment platelet over-reactivity observed by TEG system on the 5th day after admission to ICCU
  Interventions: Drug: Aspirin (200mg) and/or Plavix (150mg) dosage according to TEG
- 2 (Other): Patients who suffered acute STEMI and were treated by PPCI and recieved by Aspirin 100mg and Plavix 75mg and showed platelet inhibition observed by TEG system on the 5th day after admission to ICCU
  Interventions: Drug: Aspirin 100mg and Plavix 75mg

INTERVENTIONS:
Drug: Aspirin (200mg) and/or Plavix (150mg) dosage according to TEG — Non- responders to Aspirin or Plavix shown on TEG analysis will be treated by doubling of Aspirin (200mg) and/or Plavix (150mg) dosage
  Arms: 1
Drug: Aspirin 100mg and Plavix 75mg — Responders to standard dual antiplatelet therapy as observed by TEG analysis will continue standard doses of Aspirin and Plavix
  Arms: 2

SUMMARY:
TEG is an established technique to assess the quality of clot formation' used mainly in surgery and obstetrics to determine possible bleeding diathesis. Recently it became to be used in cardiology, where it can be a valuable tool to assess a response to antiplatelet therapy and its association with the outcome. However, there is a few data about use of TEG in STEMI patients undergoing PCI. Our study is designed to assess by TEG the platelet's response to clopidogrel treatment during acute STEMI in patients undergoing primary PCI and the correlation of this response with the long term outcome, and ability to dose adjustment according to a specific measurement by TEG in order to prevent future MACE.

DETAILED DESCRIPTION:
TEG system may provide the capabilities needed to deliver personalized therapy, first, because it can identify patients at risk of ischemic event based on hemostatic influences, particularly platelet aggregation and platelet reactivity. Secondly, because treating those patients who exhibit high platelet reactivity -- an indication that they are not reaching a therapeutic level -- with appropriate drugs and doses is expected to improve outcomes.

In this study that would be increased clopidogrel maintenance dosing (150 mg) or aspirin maintenance dosing to 200mg in an attempt to lower platelet reactivity below the 50th%ile, which we expect to also reduce their ischemic risk during the follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or more
* Patients admitted with acute STEMI as a first Coronary event
* Duration of symptoms less than 12 hours
* PCI elected as a treatment of acute STEMI
* Informed consent signed

Exclusion Criteria:

* Thrombolytic therapy
* PCI not performed after diagnostic angiography (conservative treatment, CABG)
* DES used in PPCI
* Staged PCI procedures
* Previous clopidogrel treatment at any time for any reason
* Previous myocardial infarction
* Known bleeding diathesis of any kind
* Significant renal insufficiency (GFR<40 ml/min)
* LFT disturbances (Transaminase elevation more than x3 ULN)
* Significant anemia (Hb<10) or a need for blood transfusion
* Significant Thrombocytopenia (PLT Count < 150000)
* Known Clopidogrel allergy
* Known Active peptic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
To determine usefulness of thromboelastography (TEG) as a valuable tool in assessing platelet response to clopidogrel treatment and post-treatment platelet reactivity during acute ST segment elevation myocardial infarction (STEMI). | 0ne year follow up

SECONDARY OUTCOMES:
To determine the correlation between platelet response to clopidogrel treatment and the outcome of patients who underwent percutaneous coronary intervention (PCI) for STEMI. | one year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Litovchik, MD, Principal Investigator — Assaf Harofeh MC Heart Institue; Alex Blatt, MD, Study Director — Assaf Harofeh MC ICCU Head of the Department
Locations (1):
- Assaf Harofeh MC ICCU, Zerrifin, Israel

REFERENCES:
- [Background] 1. J Am Coll Cardiol. 2007 Feb 13;49(6):657-66. Epub 2007 Jan 26. Increased risk in patients with high platelet aggregation receiving chronic clopidogrel therapy undergoing percutaneous coronary intervention: is the current antiplatelet therapy adequate? Bliden KP, DiChiara J, Tantry US, Bassi AK, Chaganti SK, Gurbel PA. 2. J Am Coll Cardiol Vol. 49, No. 14, 2007 (1505-16) Variability in Individual Responsiveness to Clopidogrel Clinical Implications, Management, and Future Perspectives Dominick J. Angiolillo, MD, PHD, FACC,* Antonio Fernandez-Ortiz, MD, PHD,† Esther Bernardo, BSC,† Fernando Alfonso, MD, PHD,† Carlos Macaya, MD, PHD,† Theodore A. Bass, MD, FACC,* Marco A. Costa, MD, PHD, FACC* 3. Circulation. 2004 Jun 29;109(25):3171-5. Epub 2004 Jun 7. Clopidogrel resistance is associated with increased risk of recurrent atherothrombotic events in patients with acute myocardial infarction. Matetzky S, Shenkman B, Guetta V, Shechter M, Bienart R, Goldenberg I, Novikov I, Pres H, Savion N, Varon D, Hod H. 4. Ann Intern Med. 2007 Mar 20;146(6):434-41. Role of clopidogrel in managing atherothrombotic cardiovascular disease. Eshaghian S, Kaul S, Amin S, Shah PK, Diamond GA. 5. Eur Heart J. 2006 Oct;27(20):2420-5. Epub 2006 Sep 27. Low response to clopidogrel is associated with cardiovascular outcome after coronary stent implantation. Geisler T, Langer H, Wydymus M, Gohring K, Zurn C, Bigalke B, Stellos K, May AE, Gawaz M. 6. Curr Pharm Des. 2006;12(10):1261-9. Clopidogrel resistance: implications for coronary stenting. Gurbel PA, Lau WC, Bliden KP, Tantry US. 7. Semin Thromb Hemost. 2007 Mar;33(2):196-202. Variable response to clopidogrel in patients with coronary artery disease. Geisler T, Gawaz M. 8. Clin Res Cardiol. 2006 Feb;95(2):122-6. Epub 2006 Jan 19. Combined aspirin and clopidogrel resistance associated with recurrent coronary stent thrombosis. Templin C, Schaefer A, Stumme B, Drexler H, von Depka M. 9. Blood Coagul Fibrinolysis. 2007 Mar;18(2):187-92. Clinical relevance of aspirin resistance in patients with stable coronary artery disease: a prospective follow-up study (PROSPECTAR). Pamukcu B, Oflaz H, Onur I, Oncul A, Ozcan M, Umman B, Mercanoglu F, Meric M, Nisanci Y. 10. Am J Cardiol. 2006 Nov 20;98(10A):11N-17N. Epub 2006 Sep 28. Aspirin resistance or variable response or both? Cheng X, Chen WH, Simon DI.